CLINICAL TRIAL: NCT04549012
Title: Tranexamic Acid Plus Oxytocin Versus Oxtocin Only in Reducing Blood Loss After Cesarean Section
Brief Title: Determination of Blood Loss After CS
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Noha Mahmoud Abu Shata, egypt, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: blood loss after CS
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Effect of Drug
MeSH Terms: interventions — Tranexamic Acid; Oxytocin

STUDY DESIGN:
Intervention Model Description: Group (A) will receive oxytocin only Group (B)will receive oxytocin plus tranexamic acid
Who Masked: Participant, Care Provider, Investigator
Masking Description: women will be given serial number ,randomization will be done through a computer generated system
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): will receive oxytocin
  Interventions: Drug: Oxytocin
- group B (Active Comparator): will receive tranexamic acid plus oxytocin
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — comparison between effect of oxytocin alone and tranexamic acid and oxytocin in reducing blood loss after CS
  Other Names: oxytocin
  Arms: group B
Drug: Oxytocin — Oxytocin
  Arms: group A

SUMMARY:
Comparing betweeen tranexamic acid plus oxytocin and oxytocin alone in their efficacy in reducing blood loss following CS

DETAILED DESCRIPTION:
tranexamic acid plus oxytocin versus oxytocin only in reducing blood loss following CS

ELIGIBILITY:
Inclusion Criteria:

1. Age : 20-40 year

   * 2- Gestational age is between 37-41weeks

3- Delivery by uncomplicated elective CS

Exclusion Criteria:

* 1- Risk factors for uterine atony such as polyhydramnios or fetal macrosomia. 2- Grandmultiparity 3- Past history of postpartum hemorrhage either atonic or traumatic 4- Previous history of retained placenta 5- Pre-eclampsia or gestational hypertension/ Maternal DM 6- Abnormal placentation 7- Contraindications to the use of tranexamic acid 8- Hypersensitivity to tranexamic acid. 9- Women receiving anticoagulant therapy. 10- having underlying disease (heart, liver, kidney, pulmonary, etc.),

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 130 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
amount of blood loss | baseline
  comparison between effect of oxytocin alone and tranexamic acid and oxytocin in reducing blood loss after CS

SECONDARY OUTCOMES:
maternal and neonatal complication | baseline
  blood transfusion ,surgical injuries ,